CLINICAL TRIAL: NCT04775355
Title: Pilot Study to Describe Changes in Urinary and Gut Microbiome During Androgen Deprivation and Radiation Therapy for Prostate Cancer
Brief Title: Study to Detect Changes in Urinary and Gut Microbiome During Androgen Deprivation Therapy and Radiation Therapy in Patients With Prostate Cancer
Status: Recruiting | Type: Observational
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 19382; NCI-2021-00700 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19382 (Other: City of Hope Comprehensive Cancer Center); P30CA033572 (NIH)
Record Dates: First submitted 2021-02-25; First posted 2021-03-01 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Stage I Prostate Cancer AJCC v7; Stage II Prostate Cancer AJCC v7; Stage IIA Prostate Cancer AJCC v7; Stage IIB Prostate Cancer AJCC v7; Stage III Prostate Cancer AJCC v7; Stage IV Prostate Cancer AJCC v7
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool, urine

GROUPS / COHORTS (1):
- Observational (biospecimen collection, questionnaire): Patients undergo collection of stool and urine samples within 2 weeks before hormone therapy or radiation therapy, after hormone therapy but before start of radiation therapy, and after completion of radiation therapy. Patients also complete a series of questionnaires prior to starting radiation therapy, mid-way through radiation therapy, and after completion of radiation therapy (within 1-3 weeks, at 3 months, and then every 6 months until 3 years from radiation completion). Patients' medical records are also reviewed.
  Interventions: Procedure: Biospecimen Collection; Other: Electronic Health Record Review; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of stool and urine
Other: Electronic Health Record Review — Medical records are reviewed
Other: Quality-of-Life Assessment — Complete quality of life questionnaires
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Complete questionnaires

SUMMARY:
This study collects urine and stool samples to determine the ability to identify changes in the microbiome (bacteria, fungi, and viruses that live in the gut and urine) of patients with prostate cancer during androgen deprivation therapy and radiation therapy. Radiation therapy has the potential to harm the genitourinary area or the bowel, causing a feeling of urgency or increased inflammation in the area. The radiation therapy is designed to not irradiate the bowel and bladder areas, but there is still some radiation exposure. The gut microbiome has been associated with differences in inflammation as well as producing molecules that influence healing. The purpose of this study is to see whether the microbiome may contribute to the healing of the organs exposed to radiation. Information learned from this study may help researchers discover a new risk factor that could be manipulated to improve the quality of life in patients with prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the feasibility of identifying changes in urine and gut microbiomes during androgen deprivation therapy and radiation therapy for prostate cancer.

SECONDARY OBJECTIVE:

I. To explore associations between baseline microbiomes and urinary or gastrointestinal radiation toxicity by Common Terminology Criteria for Adverse Events (CTCAE) and Patient Reported Outcomes (PRO).

OUTLINE:

Patients undergo collection of stool and urine samples within 2 weeks before hormone therapy or radiation therapy, after hormone therapy but before start of radiation therapy, and after completion of radiation therapy. Patients also complete a series of questionnaires prior to starting radiation therapy, mid-way through radiation therapy, and after completion of radiation therapy (within 1-3 weeks, at 3 months, and then every 6 months until 3 years from radiation completion). Patients' medical records are also reviewed.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed prostate cancer, with a plan to receive radiation therapy for either definitive (cohort A) or salvage (cohort B) therapy. Patients without planned androgen deprivation therapy (ADT) will be accrued to cohort C

  * Cohort A will be restricted to Gleason grade group 3 or higher (4+3 or 8-10) so that androgen deprivation will be indicated
  * Cohort B will not be restricted by Gleason grade but will require rising prostate-specific antigen (PSA) and a plan for ADT with salvage radiation
  * Cohort C will be prostate cancer patients in whom definitive or salvage radiation is planned without ADT
* Patients must be age 18 or older
* Willing to provide urine and stool samples at specified time points

Exclusion Criteria:

* Men with inflammatory bowel disease or pre-existing cystitis will be excluded

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with prostate cancer who are receiving definitive or salvage radiation.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-04-14 (Actual); Primary Completion 2026-07-29 (Estimated); Study Completion 2026-07-29 (Estimated)

PRIMARY OUTCOMES:
Feasibility of detecting and categorizing urinary and gut microbiota | Up to 3 years
  Will be defined as the ability to generate a microbial profile for >= 80% of samples.

SECONDARY OUTCOMES:
Detectability of changes | Up to 3 years
Detectability of associations between microbial populations and toxicity | Up to 3 years

OTHER OUTCOMES:
Changes in microbiome | Baseline up to 3 years after radiation completion
  The baseline microbiome and changes in microbiome will be evaluated for association with acute and late toxicity (graded by Common Terminology Criteria for Adverse Events) and patient reported outcomes (Functional Assessment of Cancer Therapy - Prostate [FACT-P], International Index of Erectile Function). Changes in FACT-P scores over time will be summarized as point changes (absolute value) from baseline for the first post-treatment time point and from the previous time point for all other time points. Changes in the microbiome will also be placed in context by obtaining dietary information to determine any patterns of diet which may confound or influence the changes in microbiome identified in the primary analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Tanya B Dorff, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States